CLINICAL TRIAL: NCT06446258
Title: Assessment of the Impact of Soft Tissue Mobilization on the Scar in Patients After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Piotr Ożóg, Principal Investigator, Nicolaus Copernicus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUMKscarmobilisation
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Cesarean Section Complications
Keywords: Soft tissue mobilization; Scar; Cesarean section
MeSH Terms: conditions — Cicatrix | interventions — Musculoskeletal Manipulations; Myofascial Release Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Two manual therapy treatments (myofascial release, soft tissue mobilization) in the lower abdominal area and the cesarean section scar, two weeks apart.
  Interventions: Other: Manual therapy (myofascial release, soft tissue mobilization)

INTERVENTIONS:
Other: Manual therapy (myofascial release, soft tissue mobilization) — Soft tissue mobilization will be performed by a team of experienced manual therapists.

SUMMARY:
The aim of the study is to assess the impact of soft tissue mobilization on the scar in patients after cesarean section. An additional aim is to assess the relationship between the initial stiffness and elasticity of the scar and the age of the patients, the number of cesarean sections performed, as well as the time that has passed since the last cesarean section. Two physiotherapeutic interventions will be performed in the form of mobilization of the soft tissues (myofascial release techniques) of the lower abdominal area and the cesarean section scar, two weeks apart. The researchers will perform an assessment before and after each therapeutic session, as well as 2 weeks after the last therapy (follow-up). The level of satisfaction with life (Satisfaction with Life Scale (SWLS)) as well as the area of the cesarean section scar (Vancouver Scar Scale (VSS), scar assessment according to the Mustoe classification) will be analyzed. Researchers will also assess the sequence of abdominal muscle contractions during activation of the pelvic floor muscles (ultrasound examination) and quantify the state of soft tissue tension using the MyotonPro measuring device.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-45,
* undergone at least 1 cesarean section in a period of not less than 6 months,
* not using physiotherapy for a cesarean section scar

Exclusion Criteria:

* women under 18 and over 45,
* pregnant women,
* presence of abdominal mesh,
* condition after abdominoplasty; nephrectomy; hysterectomy; cystectomy,
* uterine fibroids,
* stoma,
* occurrence of neurological symptoms (exclusion based on a functional test including the following elements: trunk flexion test in a sitting position (Slump test), Babinski test and clonic reflex test, tension tests for the sciatic nerve (passive straight leg raise test) and bowstring test and femoral nerve test (in lying on the front and on the side), examination of knee and ankle reflexes, as well as assessment of superficial sensation and strength of indicator muscles in the innervation of the lumbar-sacral spine),
* positive result of pain provocation tests: axial compression of the spine and maximum compression of the intervertebral foramen in the lumbosacral spine area,
* presence of contraindications to myofascial release therapy (active cancer, deep vein thrombosis, aneurysms, infectious diseases, viral and bacterial infections, acute inflammation and fever),
* women who underwent CC surgery in less than 6 months,
* previous surgical treatment and spine injury,
* vertical scar after cesarean section,
* use of physiotherapy treatments in the last six months,
* additionally the following comorbid conditions: cancer, diabetes, osteoporosis, diseases of the digestive system, circulatory system, rheumatic, mental and gynecological diseases, pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale (VSS) | 1. Before first intervention (baseline); 2. Before the second intervention (two weeks after the first intervention); 3. Two weeks after the second intervention (follow-up)
  The Vancouver Scar Scale (VSS) rating the scars according to four parameters: vascularity, pigmentation, pliability, and height. Each parameter contains ranked subscales that may be summed to obtain a total score ranging from 0 (representing normal skin) to 13 (representing worst scar imaginable)
Scar assessment according to the Mustoe classification | 1. Before first intervention (baseline); 2. Before the second intervention (two weeks after the first intervention); 3. Two weeks after the second intervention (follow-up)
  6-stage scar classification taking into account its shape, size, color, as well as symptoms such as pain and itching.
Satisfaction With Life Scale (SWLS) | 1. Before first intervention (baseline); 2. Before the second intervention (two weeks after the first intervention); 3. Two weeks after the second intervention (follow-up)
  The Satisfaction with Life Scale (SWLS) is used to measure the feeling of satisfaction with life. This tool consists of five statements that the respondent evaluates on a seven-point scale. The respondent assesses the extent to which each statement applies to his or her life so far. The result obtained is the overall degree of satisfaction with life. The results range from 5 to 35 points. The higher the score, the higher the sense of life satisfaction.
Assessment of the sequence of abdominal muscle contraction during activation of the pelvic floor muscles - ultrasound examination | 1. Before first intervention (baseline); 2. After first intervention; 3. Before the second intervention (two weeks after the first intervention); 4. After the second intervention; 5. Two weeks after the second intervention (follow-up)
  Sonoscape E2 device
Quantitative assessment of soft tissue tension - Stiffness (S) | 1. Before first intervention (baseline); 2. After first intervention; 3. Before the second intervention (two weeks after the first intervention); 4. After the second intervention; 5. Two weeks after the second intervention (follow-up)
  Objective parameter [N/m] quantifying the state of soft tissue tension using the MyotonPro device. Determines the force generated by the myometer's measuring tip needed to deform the tissue being examined to a specified depth. During the planned examination, the area of the cesarean section scar and the erector spinae muscle in the lumbar section will be assessed.
Quantitative assessment of soft tissue tension - Decrement (D) | 1. Before first intervention (baseline); 2. After first intervention; 3. Before the second intervention (two weeks after the first intervention); 4. After the second intervention; 5. Two weeks after the second intervention (follow-up)
  An objective parameter that quantifies the state of soft tissue tension using the MyotonPro device. It determines a property of tissue called elasticity. It is the ability of muscle tissue to return to its original shape after the deforming force ceases. During the planned examination, the area of the cesarean section scar and the erector spinae muscle in the lumbar section will be assessed.
Transversus Abdominis activation-ratio (TrA-AR) | 1. Before first intervention (baseline); 2 Before the second intervention (two weeks after the first intervention); 3. Two weeks after the second intervention (follow-up)
  Ultrasound examination (Sonoscape E2 device): TrA activation ratio is created by dividing the thickness of the transverse abdominis muscle during contraction [mm] by the thickness of the transverse abdominis muscle during resting [mm]

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Strojek, PhD, Study Chair — Department of Physiotherapy, Collegium Medicum in Bydgoszcz, Nicolaus Copernicus University in Toruń
Locations (1):
- Department of Physiotherapy, Collegium Medicum in Bydgoszcz, Nicolaus Copernicus University, Bydgoszcz, Techników 3, Poland

REFERENCES:
- [Background] Stupak A, Kondracka A, Fronczek A, Kwasniewska A. Scar Tissue after a Cesarean Section-The Management of Different Complications in Pregnant Women. Int J Environ Res Public Health. 2021 Nov 15;18(22):11998. doi: 10.3390/ijerph182211998. PMID 34831752
- [Result] Gilbert I, Gaudreault N, Gaboury I. Exploring the Effects of Standardized Soft Tissue Mobilization on the Viscoelastic Properties, Pressure Pain Thresholds, and Tactile Pressure Thresholds of the Cesarean Section Scar. J Integr Complement Med. 2022 Apr;28(4):355-362. doi: 10.1089/jicm.2021.0178. Epub 2022 Jan 13. PMID 35426735
- [Result] Li YP, Liu CL, Zhang ZJ. Feasibility of Using a Portable MyotonPRO Device to Quantify the Elastic Properties of Skeletal Muscle. Med Sci Monit. 2022 Jan 28;28:e934121. doi: 10.12659/MSM.934121. PMID 35087016
- [Result] Gilbert I, Gaudreault N, Gaboury I. Intra- and inter-evaluator reliability of the MyotonPRO for the assessment of the viscoelastic properties of caesarean section scar and unscarred skin. Skin Res Technol. 2021 May;27(3):370-375. doi: 10.1111/srt.12956. Epub 2020 Oct 21. PMID 33084197